CLINICAL TRIAL: NCT04345458
Title: Safety and Efficacy of Prefilled Liquid Etanercept(Yisaipu) for Active Ankylosing Spondylitis on the Basis of NSAID Therapy: A Multicenter Randomized, Double-blind, Parallel Group Phase III Trial
Brief Title: Safety and Efficacy Study of Prefilled Liquid Etanercept(Yisaipu) for Active Ankylosing Spondylitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sunshine Guojian Pharmaceutical (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C301S-AS III
Record Dates: First submitted 2020-04-03; First posted 2020-04-14 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Ankylosing Spondylitis
Keywords: prefilled liquid etanercept; lyophilized etanercept powder; ankylosing spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group I (Experimental): twice weekly 25 mg prefilled liquid etanercept
  Interventions: Drug: prefilled liquid etanercept(Yisaipu)
- group II (Experimental): once weekly 50 mg prefilled liquid etanercept
  Interventions: Drug: prefilled liquid etanercept(Yisaipu)
- group III (Active Comparator): 25 mg twice weekly lyophilized etanercept powder
  Interventions: Drug: lyophilized etanercept powder(Yisaipu)

INTERVENTIONS:
Drug: prefilled liquid etanercept(Yisaipu)
  Arms: group I; group II
Drug: lyophilized etanercept powder(Yisaipu)
  Arms: group III

SUMMARY:
This randomized, double-blind, phase III parallel-group non-inferiority study aimed to investigate the efficacy and safety of prefilled liquid etanercept (Yisaipu) versus lyophilized etanercept powder (Yisaipu) in active ankylosing spondylitis patients.

DETAILED DESCRIPTION:
The study carried out between March 6, 2014 and July 13, 2015 across multiple medical centers in China enrolled adult active ankylosing spondylitis patients aged between 18 and 65 years. Patients were randomized in a 3:1:1 ratio to receive twice weekly 25 mg prefilled liquid etanercept for totally 24 injections (group I) or once weekly 50 mg prefilled liquid etanercept for totally 48 injections (group II), or 25 mg twice weekly lyophilized etanercept powder for totally 48 injections (group III). The primary efficacy outcome was the proportion of patients who achieved ASAS20 at week 24.

ELIGIBILITY:
Inclusion Criteria:

* age 18-65，male or female
* Sign the informed consent
* Fulfill the 1966 AS New York criteria for axial spondyloarthritis(SpA)
* Active disease phase of SpA, defined as BASDAI≥4 or night back pain≥4 at screening
* Inadequate response to NSAID≥4 week
* Application of NSAID with stable dose for no less than 2 weeks at screening
* Stable dose of prenisone for at least four weeks at ≤10mg per day if used at screening, or stop oral use for at least 4 weeks or stop local injection at least 12 weeks
* Stable dose of any DMARD for at least four weeks if used at screening, or stop use for at least 4 weeks
* Stop and receiving washing out for at least 4 week if receiving Chinese traditional drug for AS, physical treatment, vaccication or IVIG
* Stop and receiving washing out for at least 12 week if receiving other biologics or other drug trials
* The lab exam should achieve the criteria as below
* Hb≥85g/L, 3.5×109/L≤WBC count≤10×109/L, PLT≥ lower limit of normal range, ALT≤2 fold of upper limit of normal range, serum creatine ≤upper limit of normal range. Negative pregnacy test for female patients. And promise to carry out contraception during the trial and 6 weeks after the trial is ended

Exclusion Criteria:

* Allergic condition or Allergic to IgG or any element of Yisaipu®
* Clinical or radiographic evidence of Complete ankylosis of spine
* Previous receiving TNF-a blockers therapy ≥3 months with poor response
* Achieve any following tuberculosis criteria

  1. History of active tubercolosis, or radiographic evidence of present or previous history of pulmonary tubercolosis
  2. close contact with patients with tubercolosis, or with high risk of infection of tubercolosis such as immune suppression status
  3. Strong positive of PPD skin test with diameter ≥10mm. at screen or within 3 weeks prior to screen
* Presence of acute infection or acute onset of chronic infection at screen
* Invasive fungal infection or conditional infection within 6 months prior to screen
* HBS-Ag or HBC-Ab positive at screen or history of HBS/HBC infection
* History of infection on artifitial joints
* Organ transplantation surgery within 6 months prior to screen
* Presence of other autoimmune diseases, including IBD, psoriasis, uveitis, SLE, multiple sclerosis, etc.
* History of congestive heart failure
* History of malignancies within 5 years prior to screen, excluding complete resection of squamous cell carcinoma, or basal cell carcinoma or cervical carcinoma in situ.
* AIDS or HIV infection
* History of lymphoma or lymphoproliferative disorders
* Presence of serious disorder of important organs or system
* Presence of factors which may influence the compliance

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 640 (Actual)
Dates: Start 2014-03-06 (Actual); Primary Completion 2015-07-13 (Actual); Study Completion 2015-07-20 (Actual)

PRIMARY OUTCOMES:
the proportion of patients who achieved ASAS20 | at week 24
  Axial SpondyloArthritis international Society (ASAS) ASAS20 was defined as an improvement of at least 20% in at least three of the following four domains: 1) patient global assessment VAS, 2) nocturnal back pain and total back pain VAS, 3) Bath AS Function Index (BASFI) VAS, and 4) inflammation (mean of intensity and duration of morning stiffness components from the an improvement at least one unit relative to baseline VAS score; no worsening in the remaining fourth domain.

SECONDARY OUTCOMES:
the proportion of patients who achieved ASAS40, ASAS partial remission | at weeks 12 and 24
  Axial SpondyloArthritis international Society (ASAS) ASAS40 was defined as improvement of at least 40% in at least three of the four abovementioned domains and an absolute improvement of at least two versus baseline VAS scores and no worsening versus the baseline in the remaining fourth domain. ASAS partial remission was defined as VAS scores ≤2 in each of the four abovementioned domains.
the proportion of patients who achieved ASAS 5/6 | at weeks 12 and 24
  Axial SpondyloArthritis international Society (ASAS) ASAS 5/6 was defined as an improvement of at least 20% in at least five of the following six domains: 1) C-reactive protein (CRP), and 2) spinalmobility (scoliosis) in addition to the four above mentioned domains
the proportion of patients who achieved the ASDAS clinically important and major improvement and inactive disease | at weeks 12 and 24
the proportion of patients who achieved BASDAI50 | at weeks 12 and 24
  Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) BASDAI50 was defined as a 50% or greater improvement versus the baseline BASDAI.
the proportion of patients who achieved improvement in BASDAI | at weeks 12 and 24
  It was evaluated with a 6-question questionnaire,including: 1) fatigue; 2)spinal pain; 3) pain and swelling of peripheral joints; 4) pain at entheseal sites; 5) severity of morning stiffness and 6) duration of morning stiffness by using a single-item visual analog scale (VAS), with scores ranging from 0-10 cm. After taking the answer of each question out of 10 , the BASDAI score was calculated by formula 0.2 [1+2+3+4+0.5(5+6)].
the proportion of patients who achieved improvement in BASFI | at weeks 12 and 24
  Bath AS Function Index (BASFI)
the proportion of patients who achieved improvement in BASMI scores | at weeks 12 and 24
  The Bath Ankylosing Spondylitis Metrology Index (BASMI) is a combined measure of spinal mobility and hip function.Cervical rotation, tragus-wall distance, lateral lumbar flexion( the distance of the middle fingertip moves on the side of the thigh), anterior lumbar flexion(modified schober) , intermalleolar distance were measured. And according to the measurement result, each score with 0, 1, 2 points was recorded.
the proportion of patients who achieved improvement in Maastricht Ankylosing Spondylitis Enthesitis Score (MASES) | at weeks 12 and 24
  The (MASES) index based on 13 entheses. Enthesial sites assessed include the bilateral 1st costochondral joints(L and R), 7th costochondral joints(L and R), posterior superior iliac spines(L and R), anterior superior iliac spines(L and R), iliac crests(L and R), proximal insertion of Achilles tendons(L and R), and the 5th lumbar spinous process.The score of each part with 0 or 1 points was recorded.
the proportion of patients who achieved improvement in nocturnal back pain and total back pain VAS | at weeks 12 and 24
  Nocturnal back pain and total back pain in the past week was assessed using a single-item visual analog scale (VAS), with scores ranging from 0-10 cm, where 0 represented no pain and 10 represented worst possible pain.
the proportion of patients who achieved improvement in patient global assessment and physician global assessment | at weeks 12 and 24
  Patient global assessment (PGA,disease activity rated by the patient) was recorded on a VAS from 0 to 10 cm, where 0 represented very good and 10 represented very worse. Physician global assessment (PhGA,disease activity rated by the physician) was recorded on a VAS from 0 to 10 cm, where 0 defined as no disease activity state and 10 defined as most serious disease activity state .
the proportion of patients who achieved improvement in number of swollen joints and number of tender joints | at weeks 12 and 24
the proportion of patients who achieved improvement in ESR and CRP | at weeks 12 and 24

OTHER OUTCOMES:
AEs | at weeks 2, 4, 8, 12, 16, 20 and 24
  To assesse the safety

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital clinical trial center, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhao D, He D, Bi L, Wu H, Liu Y, Wu Z, Li Y, Wang G, Li X, Bao C, Jiang L, Zhang Z, Xiao W, Tong G, Wang D, Huang F. Safety and Efficacy of Prefilled Liquid Etanercept-Biosimilar Yisaipu for Active Ankylosing Spondylitis: A Multi-Center Phase III Trial. Rheumatol Ther. 2021 Mar;8(1):361-374. doi: 10.1007/s40744-021-00276-1. Epub 2021 Feb 9. PMID 33559842